CLINICAL TRIAL: NCT00050050
Title: CBT for Residual ADHD Symptoms in Adults
Brief Title: Cognitive Behavioral Therapy for Adult Attention Deficit Hyperactivity Disorder
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Steven A. Safren, Director Behavioral Medicine, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R03MH060940 (NIH); R03MH060940 (NIH); DSIR AT-AS
Record Dates: First submitted 2002-11-20; First posted 2002-11-21 (Estimated); Last update posted 2014-05-26 (Estimated); Status verified 2014-05

CONDITIONS: Attention Deficit Disorder With Hyperactivity
Keywords: Adult; ADHD; ADD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Cognitive Behavioral Therapy; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Cognitive behavioral therapy
Drug: Drug therapy

SUMMARY:
This study will determine the effectiveness of cognitive behavioral therapy (CBT) in treating the symptoms of attention deficit hyperactivity disorder (ADHD) in adults who have not responded to drug treatment.

Study hypothesis: CBT is an effective treatment for adult ADHD.

DETAILED DESCRIPTION:
ADHD, previously believed to be a disorder of childhood, affects as many as 5 percent of adults. Adults with ADHD are at high risk for academic and occupational underachievement, relationship difficulties, and reduced quality of life. This study will determine whether CBT is more effective than drug therapy in treating ADHD symptoms in adults who have been resistant to previous drug therapies.

Participants will be randomly assigned to receive 12 to 15 weekly sessions of either CBT or drug therapy which may include new or previously taken drugs. Questionnaires will be used to assess participants' ADHD symptoms at study start and at study completion.

ELIGIBILITY:
Inclusion Criteria:

* Adult ADHD of at least moderate severity
* On current drug therapy for ADHD

Exclusion Criteria:

* Depression, panic disorder, bipolar disorder, organic mental disorders, psychotic disorders, or pervasive developmental disorders
* Current substance abuse or dependence
* IQ less than 90
* Suicide risk
* History of cognitive behavioral therapy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2001-09; Primary Completion 2003-08 (Actual); Study Completion 2003-08 (Actual)

PRIMARY OUTCOMES:
ADHD symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Steven A. Safren, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States